CLINICAL TRIAL: NCT04390750
Title: Care Partner Assisted Intervention to Improve Oral Health of Individuals With Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Duke University (Other); University of North Carolina, Chapel Hill (Other); NYU Langone Health (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-068-E; U01DE027512 (NIH)
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2023-10

CONDITIONS: Mild Dementia
Keywords: oral health; oral hygiene; dementia; care partner; periodontal disease
MeSH Terms: conditions — Dementia; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: 3 Groups - 2 Treatment Groups, 1 Control Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group 1 (No Intervention): Treatment Group 1 will receive a standard educational booklet, a clinical oral health evaluation and a smart electronic toothbrush with no instruction on oral hygiene technique. The study coordinator will download the toothbrush data for data collection. The dental hygienist will observe the participant's normal toothbrushing technique, interdental cleaning procedures and the cleaning of partial dentures. No instruction is provided. The hygienist will provide basic instruction on proper use of the smart electronic toothbrush.
- Treatment Group 2 (Experimental): Treatment Group 2 will receive a standard educational booklet, a smart electronic toothbrush, a clinical oral health evaluation with tailored instruction on oral hygiene technique and care partner coaching. The study coordinator will download the toothbrush data for data collection. The dental hygienist and interventionist will work together to fulfill the following intervention components: tailored instruction and coaching.
  Interventions: Behavioral: Care Partner-Assisted Intervention
- Control Group (No Intervention): The Control group will receive a standard educational booklet and a clinical oral health evaluation with no instruction on oral hygiene technique. The dental hygienist will observe the participant's normal toothbrushing technique, interdental cleaning procedures and the cleaning of partial dentures. No instruction is provided.

INTERVENTIONS:
Behavioral: Care Partner-Assisted Intervention — Tailored teaching and coaching
  Arms: Treatment Group 2

SUMMARY:
Care Partner Assisted Intervention to Improve Oral Health for Individuals with Mild Dementia is a randomized control trial (RCT) based in New York City and North Carolina. The intervention includes both a tailored oral care plan and a behavioral component using the Adaptive Leadership Framework for Chronic Illness that the team introduced to manage symptoms associated with chronic conditions, such as dementia. Objective 1 is to evaluate the efficacy of an intervention to improve oral hygiene clinical outcomes (i.e. plaque index and gingival index) by improving oral hygiene behavior (i.e., frequency and duration of toothbrushing) and oral health skills among individuals with mild dementia. Objective 2A is to determine whether effects of the intervention on oral hygiene behavioral outcomes, are mediated by the following variables from the care partners' perspective: 1) oral care self-efficacy; 2) care partner self-efficacy; 3) use of cueing methods; 4) and FOCUSED Communication. Objective 2B is to determine whether effects of the intervention on oral hygiene clinical outcomes, are mediated by the following variables from the care partner's perspective: 1) oral care self-efficacy; 2) care partner's self-efficacy; 3) use of cueing methods; 4) and FOCUSED Communication. Objective 3A is to determine whether effects of the intervention on oral hygiene clinical outcomes are mediated by oral hygiene behavioral outcomes. Objective 3B is to determine whether effects of the intervention on oral hygiene clinical outcomes are mediated by the care partner's factors, which then mediate the oral hygiene behavioral outcomes on oral hygiene clinical outcomes. This innovative care partner-assisted oral care behavior intervention will assist participants and care partners in implementing a cooperative oral hygiene care plan to prevent deterioration of oral health, which in turn, will help the targeted population maintain independence in completing daily activities and quality of life for an extended period of time.

DETAILED DESCRIPTION:
Dyads that each consist of an individual with mild dementia and his/her care partner will be enrolled at two sites, Duke University in Durham, North Carolina and New York University in New York, New York. This is an unblinded, randomized trial to assess the acceptability and effectiveness of the oral health intervention among individuals with mild dementia (MD). The study will utilize qualitative and quantitative methods to learn about the oral health outcomes in individuals with mild dementia.

The study lasts 6 months. The first three months is the active intervention phase in which coaching and educational modules are delivered. The second three months is the maintenance period in which no coaching or educational modules are presented to participants. As a team, the study coordinator, the oral health evaluator (a dental hygienist), and the interventionist will conduct three visits with the participants and their care partners; baseline, 3-month (end of the active intervention phase), and 6-month (end of three-month maintenance phase).

The intervention protocol will include three groups; two treatment groups and one control group. All participants will receive oral health education material at the baseline visit. Treatment Group 1 and Treatment Group 2 will be given a smart electronic toothbrush. Only Treatment Group 2 will receive the in-home and telephone coaching throughout the duration of the study and will be instructed to record daily brushing habits. The coaching sessions include individualized instruction on oral hygiene technique, cueing strategy development, or oral hygiene monitoring and coaching. Treatment Group 1 and the Control Group will not receive the coaching sessions.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of mild dementia
* have at least 4 natural teeth
* 60 years and older
* living with an informal caregiver (i.e. care partner) who is age 18 or older and is willing to participate in the intervention
* community-dwelling and physically able to brush own teeth
* We will use the following guidelines to identify those with mild dementia: a) a diagnosis of dementia by a physician with dementia expertise within the past year, b) from medical records, a recent Montreal Cognitive Assessment (MoCA) score > 14 or a Mini-Mental Status Examination (MMSE) score > 16, and c) can follow 2 to 3-step commands

Exclusion Criteria:

* unable to have an oral health evaluation
* prescribed antibiotics prior to a regular dental visit
* has sensory or physical problems that prevent participation in the intervention
* has a terminal illness or behavioral or psychiatric disorder that would interfere with participation in the intervention
* has a medical condition such as serious congenital heart conditions, previous infective endocarditis, prosthetic cardiac valves, and cardiac transplantation with cardiac valvulopathy that places him/her at greater risk of infection from the manipulation of the gums to measure the gingival index
* has a medical condition that suppresses the immune system
* has had a total joint replacement and has had an infection in the replaced joint
* is at increased risk of bleeding due to bleeding disorder such as hemophilia or the use of anti-platelet therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bei Wu, PhD, Principal Investigator — New York University
Locations (2):
- United States (2):
  - New York City (Participants Homes), New York, New York
  - North Carolina (Participants Homes), Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be shared between 9 months and 36 months following article publication or as required by a condition of awards and agreements supporting the research, for researchers who provide a methodologically sound proposal. Data will be made available at https://www.icpsr.umich.edu/web/pages (Note: a specific link will be provided after the study is published/when the DOI is obtained.) The protocol, statistical analysis plan, and analytic code will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Data will be made available at Clinicaltrials.gov and ICPSR (a specific link will be provided after the study is published/when the DOI is obtained).

REFERENCES:
- [Derived] Wu B, Plassman BL, Poole P, Siamdoust S, Bunn M, Burwell B, Pei Y, Downey C, Gomes D, Kamer A, Yu G, Leak Bryant A, Anderson RA. Study protocol for a randomised controlled trial of a care partner assisted intervention to improve oral health of individuals with mild dementia. BMJ Open. 2022 Jun 22;12(6):e057099. doi: 10.1136/bmjopen-2021-057099. PMID 35732396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the NYU ADRC, Duke Memory Disorders Clinic, and Montefiore CEAD. At NYU and CEAD, potential participants were identified from upcoming appointments, informed about the study by staff, and screened by phone. CEAD collaborators also partnered with community organizations to reach diverse populations. At Duke, participants were identified via electronic medical records, sent a letter, and contacted by a coordinator for phone screening.
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Started | 20 | 20 | 20
Completed | 18 | 17 | 19
Not Completed | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.05 (6.61) | 74.65 (6.43) | 76.35 (6.77) | 75.35 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 10 | 27
  Male | 11 | 12 | 10 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Hispanic | 2 | 1 | 1 | 4
  Race/ethnicity: Non-Hispanic Black | 3 | 4 | 4 | 11
  Race/ethnicity: Non-Hispanic White | 15 | 15 | 15 | 45
Plaque Index [Mean (Standard Deviation); unit: Proportion of sites with plaque deposits] — UNC Modified Green and Vermillion Oral Hygiene Index. The index value is the proportion of sites with plaque deposits.
  Proportion of sites with plaque deposits | 0.62 (0.32) | 0.60 (0.25) | 0.54 (0.32) | 0.59 (0.31)
Gingival Index [Mean (Standard Deviation); unit: Proportion of sites with inflammation] — UNC Modified Loe and Silness Gingival Index. The index value is the proportion of sites with inflammation.
  Proportion of sites with inflammation | 0.68 (0.34) | 0.59 (0.38) | 0.52 (0.37) | 0.60 (0.36)
Frequency of Toothbrushing [Count of Participants; unit: Participants]
  < Twice a day | 7 | 8 | 7 | 22
  >= Twice a day | 13 | 12 | 13 | 38
Duration of Toothbrushing [Count of Participants; unit: Participants]
  >= 2 minutes | 5 | 6 | 7 | 18
  >= 1 min & < 2 minutes | 8 | 11 | 7 | 26
  < 1 minute | 7 | 3 | 6 | 16
Frequency of interdental cleaning [Count of Participants; unit: Participants]
  Twice a day or more | 7 | 4 | 5 | 16
  Once a day | 4 | 4 | 4 | 12
  Several times a week | 2 | 2 | 3 | 7
  Once or less than once a week | 1 | 4 | 2 | 7
  Hardly ever | 1 | 3 | 4 | 8
  Never | 4 | 3 | 2 | 9
  Unknown | 1 | 0 | 0 | 1
Interproximal cleaning technique [Count of Participants; unit: Participants]
  Less than optimal | 18 | 15 | 12 | 45
  Optimal | 2 | 5 | 8 | 15
Oral health knowledge score [Mean (Standard Deviation); unit: Scores on a scale] | 0.66 (0.19) | 0.65 (0.18) | 0.68 (0.15) | 0.66 (0.18)
Oral health hygiene score [Mean (Standard Deviation); unit: Scores on a scale] | 2.18 (0.41) | 1.88 (0.43) | 1.82 (0.53) | 1.96 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: UNC Modified Green and Vermillion Oral Hygiene Index. Plaque was measured per tooth, 0 = No plaque, 1 = Plaque covers <1/3 tooth, 2 = Plaque covers >=1/3 but <2/3 tooth and 3 = Plaque covers >=2/3 tooth. The index values were calculated as the proportion of sites with plaque deposits on at least less than 1/3 of crown. The index value is the proportion of sites with plaque deposits. Higher index values indicate higher levels of plaque.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Mean (Standard Deviation); unit: Proportion of sites with plaque deposits
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Proportion of sites with plaque deposits | 0.55 (0.36) | 0.41 (0.25) | 0.48 (0.32)
Statistical Analysis 1: Comparison: Treatment Group 1 vs Control Group; A linear mixed effects model including an arm-by-time interaction was used to estimate between-arm differences in change in plaque levels at the primary endpoint of 3 months; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on plaque levels between Treatment Group 1 and Control at 3 months; p = 0.939, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = 0.00, 95% CI 2-sided [-0.11 to 0.11]
Statistical Analysis 2: Comparison: Treatment Group 2 vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on plaque levels between Treatment Group 2 and Control at 3 months; p = 0.103, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = -0.09, 95% CI 2-sided [-0.21 to 0.02]

2. Primary Outcome: Gingival Index
Description: UNC Modified Loe and Silness Gingival Index Gingival inflammation is evaluated per tooth, classified as 0 = Normal gingiva, 1 = Mild inflammation, no bleeding on probing, 2 = Moderate inflammation, bleeding on probing, 3 = Severe inflammation, tendency to spontaneous bleeding. Index values were calculated as the proportion of sites with at least some mild inflammation. The index value is the proportion of sites with inflammation. Higher index values indicate greater gingival inflammation.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Mean (Standard Deviation); unit: Proportion of sites with inflammation.
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Proportion of sites with inflammation. | 0.61 (0.39) | 0.37 (0.39) | 0.47 (0.42)
Statistical Analysis 1: Comparison: Treatment Group 1 vs Control Group; A linear mixed effects model including an arm-by-time interaction was used to estimate between-arm differences in change in gingival inflammation at the primary endpoint of 3 months; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on gingival inflammation between Treatment Group 1 and Control at 3 months; p = 0.995, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = 0.00, 95% CI [-0.16 to 0.16]
Statistical Analysis 2: Comparison: Treatment Group 2 vs Control Group; [analysis description as in outcome 2, analysis 1]; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on gingival inflammation between Treatment Group 2 and Control at 3 months; p = 0.132, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = -0.12, 95% CI [-0.28 to 0.04]

3. Primary Outcome: Plaque Index
Description: as for outcome 1
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Mean (Standard Deviation); unit: Proportion of sites with plaque deposits
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Proportion of sites with plaque deposits | 0.55 (0.35) | 0.45 (0.28) | 0.53 (0.30)
Statistical Analysis 1: Comparison: Treatment Group 1 vs Control Group; A linear mixed effects model including an arm-by-time interaction was used to estimate between-arm differences in change in plaque levels at the secondary endpoint of 6 months; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on plaque levels between Treatment Group 1 and Control at 6 months; p = 0.402, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = -0.05, 95% CI 2-sided [-0.16 to 0.06]
Statistical Analysis 2: Comparison: Treatment Group 2 vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on plaque levels between Treatment Group 2 and Control at 6 months; p = 0.072, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = -0.10, 95% CI 2-sided [-0.21 to 0.01]

4. Primary Outcome: Gingival Index
Description: as for outcome 2
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Mean (Standard Deviation); unit: Proportion of sites with inflammation.
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Proportion of sites with inflammation. | 0.58 (0.39) | 0.43 (0.35) | 0.63 (0.41)
Statistical Analysis 1: Comparison: Treatment Group 1 vs Control Group; A linear mixed effects model including an arm-by-time interaction was used to estimate between-arm differences in change in gingival inflammation at the secondary endpoint of 6 months; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on gingival inflammation between Treatment Group 1 and Control at 6 months; p = 0.014, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = -0.20, 95% CI 2-sided [-0.36 to -0.04]
Statistical Analysis 2: Comparison: Treatment Group 2 vs Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Other — The effect estimate reflects the adjusted difference in change from baseline on gingival inflammation between Treatment Group 2 and Control at 6 months; p = 0.005, Linear mixed effects model; Linear mixed effects model with arm-by-time interaction; Interaction coefficient = -0.23, 95% CI 2-sided [-0.39 to -0.07]

5. Secondary Outcome: Frequency of Toothbrushing
Description: Participants' frequency toothbrushing Categorical variable with the following response types: 'Less than Twice a Day' or 'Twice a Day or more'.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Participants
  < Twice a week | 2 | 4 | 6
  >= Twice a week | 16 | 13 | 12

6. Secondary Outcome: Frequency of Toothbrushing
Description: as for outcome 5
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Participants
  < Twice a week | 3 | 4 | 4
  >= Twice a week | 15 | 13 | 15

7. Secondary Outcome: Duration of Toothbrushing
Description: Participants' duration of toothbrushing. Reported by the dental hygienist. Categorical variable consisting of 3 response types (< 1minute; > 1 minute & < 2minute; > 2 minute per toothbrushing session).
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Participants
  >= 2 min | 10 | 9 | 4
  >= 1 min & < 2 min | 5 | 6 | 8
  < 1min | 3 | 1 | 6
  Unknown | 0 | 1 | 0

8. Secondary Outcome: Duration of Toothbrushing
Description: as for outcome 7
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Participants
  >= 2 min | 5 | 8 | 6
  >= 1 min & < 2 min | 10 | 7 | 9
  < 1min | 3 | 2 | 4
  Unknown | 0 | 0 | 0

9. Secondary Outcome: Frequency of Interdental Cleaning
Description: Participants' frequency of interdental cleaning Collected via self-report via care partner. Categorical variable ranging from 'Never' to 'Twice a Day or More'.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Participants
  Twice a day or more | 4 | 4 | 5
  Once a day | 6 | 4 | 3
  Several times a week | 3 | 2 | 3
  Once or less than once a week | 1 | 5 | 4
  Hardly ever | 0 | 1 | 1
  Never | 4 | 1 | 2

10. Secondary Outcome: Frequency of Interdental Cleaning
Description: Participants' frequency of interdental cleaning. Collected via self-report via care partner. Categorical variable ranging from 'Never' to 'Twice a Day or More'.
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Participants
  Twice a day or more | 4 | 4 | 5
  Once a day | 4 | 4 | 7
  Several times a week | 5 | 2 | 1
  Once or less than once a week | 0 | 3 | 1
  Hardly ever | 3 | 2 | 2
  Never | 2 | 2 | 3

11. Secondary Outcome: Interproximal Cleaning Technique
Description: Participants' Interproximal Cleaning Technique Reported by the dental hygienist. Categorical variable, with the following response types: 'Less than Optimal' or 'Interproximal Surfaces Cleaned Using 'C' shape'.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Participants
  Less than optimal | 14 | 11 | 10
  Optimal | 4 | 6 | 8

12. Secondary Outcome: Interproximal Cleaning Technique
Description: Participants' Interproximal Cleaning Technique. Reported by the dental hygienist. Categorical variable, with the following response types: 'Less than Optimal' or 'Interproximal Surfaces Cleaned Using 'C' shape'.
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Participants
  Less than optimal | 13 | 9 | 11
  Optimal | 5 | 8 | 8

13. Secondary Outcome: Oral Health Hygiene Score
Description: Participant Oral Hygiene Skills. Reported by the dental hygienist. Average score on the Oral Hygiene Assessment Sheet of Routine Care Questionnaire. Scores range from 1 to 3. Lower scores indicate higher oral health hygiene.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Scores on a scale | 1.83 (0.67) | 1.64 (0.44) | 1.78 (0.45)

14. Secondary Outcome: Oral Health Hygiene Score
Description: Participant Oral Hygiene Skills. Reported from dental hygienist. Average score on the Oral Hygiene Assessment Sheet of Routine Care Questionnaire. Scores on this scale range from 1 to 3. Lower scores indicate higher oral health hygiene.
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Scores on a scale | 1.85 (0.53) | 1.58 (0.46) | 1.85 (0.43)

15. Secondary Outcome: Oral Health Knowledge Score
Description: Participant Oral Health Knowledge Score Scores were calculated as the proportion of correct responses on the Modified Oral Health Knowledge section of the Study Participant Questionnaire. Higher scores indicate greater oral health knowledge. Range is 0-1.
Time Frame: 3 months
Population: 6 participants were withdrawn after the baseline visit, and 1 participant did not complete assessment at 3 months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 18
Scores on a scale | 0.71 (0.20) | 0.81 (0.12) | 0.73 (0.17)

16. Secondary Outcome: Oral Health Knowledge Score
Description: as for outcome 15
Time Frame: 6 months
Population: 6 participants were withdrawn after the baseline visit.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
Number analyzed (Participants) | 18 | 17 | 19
Scores on a scale | 0.65 (0.24) | 0.76 (0.19) | 0.68 (0.15)

ADVERSE EVENTS:
Time Frame: Up to 6 months from Enrollment Date
Description: Subjects were monitored for adverse events over a 6-month period, beginning at enrollment and continuing through the last study visit.
Arm/Group | Treatment Group 1 | Treatment Group 2 | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group 1 (N=20) | Treatment Group 2 (N=20) | Control Group (N=20)
Gum Soreness (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Tissue Trauma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
We were unable to meet target accrual which may have limited the ability to detect statistically significant differences across arms, primarily due to the following barriers: reduced frequency of patient visits to clinics during the COVID-19 pandemic, which limited in-person recruitment and establishing relationships with non-affiliated hospitals and organizations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04390750/Prot_SAP_000.pdf